CLINICAL TRIAL: NCT07181395
Title: Comparison of the Effectiveness of Two Different Mulligan Mobilization Techniques in Patients With Non-Specific Low Back Pain: A Triple-Blind Randomized Controlled Trial
Brief Title: Mulligan Mobilization Techniques for Non-Specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Bulent ELBASAN, Professor Dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GU-ETHICS-2025-08-863; GU-Ethics-08/863 (Other: Gazi University Ethics Committee)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-specific Low Back Pain (NSLBP)
Keywords: Mulligan Mobilization, Hip Internal Rotation, Straight Leg Raise, Physiotherapy, Manual Therapy, Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a triple-blind study. Participants, outcome assessors, and investigators performing data analysis are blinded to group allocation. Only physiotherapists delivering the interventions are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy + Hip Internal Rotation Mulligan Mobilization (Experimental): Participants will receive conventional physiotherapy combined with Mulligan mobilization applied to hip internal rotation. The mobilization will be performed with a mobilization belt, 3 sets of 10 repetitions, twice weekly for 4 weeks.
  Interventions: Behavioral: Hip Internal Rotation Mulligan Mobilization; Behavioral: Conventional Physiotherapy
- Conventional Physiotherapy + Straight Leg Raise Mulligan Mobilization (Experimental): Participants will receive conventional physiotherapy combined with Mulligan mobilization applied to straight leg raise under traction. The mobilization will be performed in 3 sets of 10 repetitions (15-20 seconds hold), twice weekly for 4 weeks.
  Interventions: Behavioral: Straight Leg Raise Mulligan Mobilization; Behavioral: Conventional Physiotherapy
- Conventional Physiotherapy Only (Active Comparator): Participants will receive conventional physiotherapy only, including transcutaneous electrical nerve stimulation (20 minutes), massage, stretching and strengthening exercises for lumbar muscles, postural training, and patient education. Treatment will be delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Conventional Physiotherapy

INTERVENTIONS:
Behavioral: Hip Internal Rotation Mulligan Mobilization — Mulligan mobilization applied to hip internal rotation using a mobilization belt. Performed in 3 sets of 10 repetitions, twice weekly for 4 weeks, in addition to conventional physiotherapy.
  Other Names: Mulligan Hip IR Mobilization
  Arms: Conventional Physiotherapy + Hip Internal Rotation Mulligan Mobilization
Behavioral: Straight Leg Raise Mulligan Mobilization — Mulligan mobilization applied to straight leg raise under manual traction. Performed in 3 sets of 10 repetitions (15-20 seconds hold), twice weekly for 4 weeks, in addition to conventional physiotherapy.
  Other Names: Mulligan SLR Mobilization
  Arms: Conventional Physiotherapy + Straight Leg Raise Mulligan Mobilization
Behavioral: Conventional Physiotherapy — Conventional physiotherapy including transcutaneous electrical nerve stimulation (20 minutes), massage, lumbar stretching and strengthening exercises, postural training, and patient education. Delivered twice weekly for 4 weeks.
  Other Names: Standard Physiotherapy

SUMMARY:
This study aims to compare the effectiveness of two different Mulligan mobilization techniques in patients with non-specific low back pain. A total of 30 adults with chronic low back pain will be randomly assigned to three groups: (1) conventional physiotherapy plus hip internal rotation Mulligan mobilization, (2) conventional physiotherapy plus straight leg raise Mulligan mobilization, or (3) conventional physiotherapy only. The interventions will be applied twice a week for four weeks. The main outcomes are pain intensity (measured by Visual Analog Scale) and lumbar range of motion. Secondary outcomes include disability level (Oswestry Disability Index) and back awareness (Fremantle Back Awareness Questionnaire). The study will help determine whether Mulligan techniques provide additional benefits beyond conventional physiotherapy in reducing pain and improving function in people with non-specific low back pain.

DETAILED DESCRIPTION:
Low back pain is the second most common cause of disability worldwide and significantly affects quality of life and healthcare systems. Non-specific low back pain (NSLBP) accounts for nearly 85% of all low back pain cases and is associated with loss of function, reduced productivity, and psychological problems. Physiotherapy approaches such as exercise, manual therapy, electrotherapy, and patient education are widely used, but not all patients benefit equally, highlighting the need for innovative and individualized treatment strategies. Mulligan mobilization is a manual therapy method that combines physiological joint movements with pain-free mobilization techniques. Techniques such as hip mobilization and traction-assisted straight leg raise (SLR) are thought to improve pain, range of motion, and functional outcomes. Although some studies suggest positive effects of Mulligan techniques, there is a lack of randomized controlled trials directly comparing different Mulligan approaches in patients with NSLBP. This triple-blind randomized controlled trial will investigate the comparative effectiveness of two Mulligan mobilization techniques. Thirty adults with NSLBP will be randomly assigned into three groups: (1) conventional physiotherapy plus hip internal rotation Mulligan mobilization, (2) conventional physiotherapy plus SLR Mulligan mobilization, and (3) conventional physiotherapy only. Interventions will be delivered twice a week for four weeks by experienced physiotherapists certified in the Mulligan Concept®. The primary outcomes will be pain intensity measured with the Visual Analog Scale (VAS) and lumbar range of motion assessed by goniometer. Secondary outcomes include disability level measured with the Oswestry Disability Index (ODI) and back awareness assessed with the Fremantle Back Awareness Questionnaire (FreBAQ). The findings of this study are expected to provide evidence on whether Mulligan mobilization techniques offer additional benefits beyond conventional physiotherapy in the management of non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with non-specific low back pain (NSLBP) for at least 3 months
* Able to walk independently
* Willing to participate and provide written informed consent

Exclusion Criteria:

* Specific causes of low back pain (e.g., disc herniation, spinal stenosis, tumor)
* Presence of neurological deficits or radiculopathy
* Hip joint pathologies limiting mobility (e.g., osteoarthritis)
* History of lumbar surgery in the last 6 months
* Diagnosed osteoporosis or osteopenia
* Contraindications for Mulligan mobilization
* Severe physical or cognitive impairments preventing participation
* Participation in other physiotherapy or manual therapy treatments during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2025-10-07 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale, VAS) | Baseline (week 0) and post-treatment (week 4).
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 100 mm horizontal line ranging from "no pain" to "worst pain imaginable." Participants will mark their pain level, and the distance in millimeters will be recorded.
Lumbar Range of Motion (ROM) | Baseline (week 0) and post-treatment (week 4).
  Lumbar spinal range of motion will be measured using a goniometer. Participants will perform active forward flexion, and the angle of motion will be recorded in degrees.

SECONDARY OUTCOMES:
Disability Level (Oswestry Disability Index - ODI) | Baseline (week 0) and post-treatment (week 4)
  Functional disability will be assessed using the Oswestry Disability Index (ODI). The scale consists of 10 items, each scored from 0 to 5, with higher scores indicating greater disability. The total score ranges from 0 (no disability) to 50 (maximum disability).
Back Awareness (Fremantle Back Awareness Questionnaire - FreBAQ) | Baseline (week 0) and post-treatment (week 4).
  Body perception related to the lumbar region will be measured using the Fremantle Back Awareness Questionnaire (FreBAQ). The questionnaire has 9 items scored on a Likert scale (0-4), with higher scores reflecting reduced back awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No